CLINICAL TRIAL: NCT07313046
Title: THE EFFECT OF TRAİNİNG PROVİDED TO CAREGİVERS ON PREVENTİNG PRESSURE ULCERS İN PATİENTS RECEİVİNG HOME CARE SERVİCES
Brief Title: CAREGİVER TRAİNİNG AND PRESSURE ULCER PREVENTİON İN HOME CARE
Acronym: CARE-PU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Perihan ARAÇLIOĞLU, LEAD INVESTIGATOR, Bartın Unıversity
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-SBB-0615
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pressure Ulcer Prevention; Pressure Ulcer Prevention Training for Home Care Patients
Keywords: pressure ulcer, prevention, home care, caregiver training
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregiver Training Intervention (Experimental): In this section, a structured training program aimed at preventing pressure ulcers will be implemented for individuals providing care to patients receiving home care services. The training program covers pressure ulcer risk factors, skin assessment, repositioning techniques, care approaches to reduce pressure, and basic skin care. The training aims to improve caregivers' knowledge and care practices.
  Interventions: Behavioral: Caregiver Training Program

INTERVENTIONS:
Behavioral: Caregiver Training Program — A structured education program for caregivers about pressure ulcer risk factors, skin care, repositioning, and care practices for pressure reduction.

SUMMARY:
Pressure ulcers are a significant health problem commonly seen in home care patients who are bedridden or have limited mobility, negatively affecting their quality of life. The knowledge and skills of caregivers play a crucial role in preventing these ulcers.

This study aims to examine whether training provided to caregivers of patients receiving home care reduces the risk of pressure ulcer formation. As part of the study, caregivers will receive training on pressure ulcer risk factors, skin care, repositioning, pressure protection methods, and appropriate care practices.

The pressure ulcer risk levels of patients will be assessed before and after the training, and the effect of the training will be compared. The results are expected to contribute to the development of caregiver training in home care services and the prevention of pressure ulcers.

DETAILED DESCRIPTION:
Pressure ulcers are a common health problem among patients receiving home care services and experiencing limited mobility. They are preventable but can lead to serious consequences. Prolonged pressure, compromised skin integrity, malnutrition, and inadequate care practices play a significant role in the development of these ulcers. The knowledge and skill level of caregivers providing care to patients in the home environment is a decisive factor in preventing pressure ulcers.

This study was designed to evaluate the effect of training provided to caregivers of patients receiving home care services on the risk of pressure ulcer development in patients. Patients receiving home care services who are at risk of pressure ulcers and the individuals providing care to these patients will be included in the study.

The training program for caregivers will cover pressure ulcer risk factors, skin assessment, repositioning frequency, pressure-reducing practices, hygiene, and basic skin care. The training will be delivered using structured training materials.

Within the scope of the study, the risk of pressure ulcers in patients will be measured using an appropriate risk assessment scale before and after the training. The findings aim to reveal the role of caregiver training in the prevention of pressure ulcers in home care services.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

The study includes:

* Patients registered with the Home Care Health Unit,
* Volunteers willing to participate in the study,
* Caregivers of patients classified as high or medium risk according to the Braden Risk Assessment Scale,
* • Caring for a patient who is not cared for by different individuals,
* Aged 18 years or older,
* Able to speak Turkish,
* Without speech or hearing problems,
* Cognitive competence sufficient to understand and answer questions.

Exclusion Criteria:

* • Not registered with the Home Care Health Unit,

  * Whose patient is classified as low risk according to the Braden Risk Assessment Scale,
  * • Those with more than one caregiver,
  * Those who did not agree to participate in the study,
  * Those under the age of 18,
  * Those who did not speak Turkish,
  * Those with speech and hearing problems,
  * Caregivers who did not have the cognitive ability to understand and answer the questions were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Pressure Ulcer Risk Level | Baseline and 4 weeks after training
  The pressure ulcer risk level of home care patients will be assessed before and after the caregiver training using a validated pressure ulcer risk assessment tool.
Pressure Ulcer Risk Level | Baseline and 3 weeks after training
  The risk level of pressure ulcer development in patients receiving home care services will be measured using a valid risk assessment tool before and after the training provided to caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Karahan, PhD, Study Director — Bartın Unıversity; Sevim ÇELİK, PhD, Study Director — Bartın Unıversity; Sibel ALTINTAŞ, PhD, Study Director — Bartın Unıversity
Locations (1):
- Bartın University, Bartın, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality considerations.

REFERENCES:
- [Background] Afzali Borojeny L, Albatineh AN, Hasanpour Dehkordi A, Ghanei Gheshlagh R. The Incidence of Pressure Ulcers and its Associations in Different Wards of the Hospital: A Systematic Review and Meta-Analysis. Int J Prev Med. 2020 Oct 5;11:171. doi: 10.4103/ijpvm.IJPVM_182_19. eCollection 2020. PMID 33312480